CLINICAL TRIAL: NCT07060976
Title: Evaluation of Dermatological Safety of Test Products by 24 Hours Patch Test Under Complete Occlusion | Semi Occlusion |Open Patch on Adult Healthy Human Subjects
Brief Title: To Check Dermatological Safety of Test Products by 24 Hours Patch Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novamed Laboratories Pvt. Ltd. (Industry)
Collaborators: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB250023-NL
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Gene Expression; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Each participant will receive Transdermal patches on the back, including the test product(s), a negative control (0.9% Saline), and a positive control (1% sodium lauryl sulfate). Reactions will be assessed at specified time intervals using a standardized Draize Scale
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): 18 Transdermal patches along with positive and negative controls
  1. Capsaicin0.025% Topical Patch,
  2. Diclofenac Diethylamine 100mg Transdermal Patch,
  3. Diclofenac Diethylamine 200mg Transdermal Patch,
  4. Diclofenac Sodium 140 mg Gel Patch,
  5. Ketoprofen20 mgTransdermalPatch,
  6. Ketoprofen30 mg Transdermal Patch,
  7. Lidocaine& Menthol Topical Patch,
  8. Lidocaine350 mg Topical Patch,
  9. Lidocaine 4% Topical Patch,
  10. Menthol 1.25% Camphor3% Capsaicin 0.025% Topical Patch,
  11. Menthol 1.25% Capsaicin0.025% Topical Patch,
  12. Menthol10% Topical Patch,
  13. Menthol5% Hydrogel Patch,
  14. Menthol 5% Topical Patch,
  15. Menthol6.0% Camphor3.1% MethylSalicylate 10%,
  16. Menthol 6.5% Topical Patch,
  17. Menthol7% Camphor 7%Topical Patch,
  18. Menthol7.5% 1×1 cm of each Patch (1 cm2) will be applied on subject's back along with 1% SLS (Positive control) and 0.9% Normal saline (Negative Control)
  Interventions: Other: 18 Transdermal patches along with positive and negative controls 1)Capsaicin0.025% Topical Patch, 2)Diclofenac Diethylamine 100mg Transdermal Patch, 3)Diclofenac Diethylamine 200mg Transdermal Patch,

INTERVENTIONS:
Other: 18 Transdermal patches along with positive and negative controls 1)Capsaicin0.025% Topical Patch, 2)Diclofenac Diethylamine 100mg Transdermal Patch, 3)Diclofenac Diethylamine 200mg Transdermal Patch, — Dose: 1×1 cm of each Patch (1 cm2) Route of administration: Topical Mode of usage: Products will be evaluated through the complete occlusion for 24 hours. At 24 hours post-application, patches will be removed and skin will be evaluated for irritation reactions at 30 mins,24 hours (Day 1)post patch removal and 168 hours (Day 7) post-patch removal (if needed). Frequency: single application

SUMMARY:
To Check Dermatological Safety of Test Products by 24 Hours Patch Testing

DETAILED DESCRIPTION:
This is single center, evaluator-blinded study in healthy adult human subjects. Single 24-hour application of sponsor(s) provided test products along with positive and negative controls will be kept in contact with the skin of subjects under occlusion |Semi occlusion |Open patch for at least 24 hours (+ 2 hours). Study can be conducted in multiple groups. Safety will be assessed throughout the study by monitoring of adverse events.

Subject's back i.e. between the scapula and waist will be utilized as application sites. Application sites will be evaluated for scoring the reaction, namely, erythema, dryness, and wrinkles on a 0-4 point scale separately for each parameter and oedema on another 0-4 points scale as per the Draize Scale after 30+5 minutes of patch removal, 24±2 hours and 168±2 hours after patch removal.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Subject with normal Fitzpatrick skin type III to V (Human skin colour determination scale).
4. Females of childbearing potential must have a self-reported negative pregnancy test.
5. Subject who do not have any previous history of adverse skin conditions and are not under any medication likely to interfere with the results.
6. Subject is in good general health as determined by the Investigator on the basis of medical history.
7. Subjects is willing to maintain the test patches in designated positions for 24 Hours.
8. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
9. Subject must be able to understand and provide written informed consent to participate in the study.
10. Subject is willing to refrain from vigorous physical exercise during the study period and follow all the instruction given.
11. For Sensitive Specific Skin Study Only:

    * Subject scoring greater than 30 for Section 2 - Sensitive v/s Resistant skin in modified Dr Baumann's* skin type questionnaire.
    * Subject with sensitive skin as confirmed by Lactic Acid Stinging Test.

Exclusion Criteria:

1. Subject having skin irritation, blemishes, excessive hair, moles, pigmentation, pimples, marks (e.g. tattoos (within the previous 3 months), scars, sunburn), open wounds, cuts, abrasions, irritation symptoms or any dermatological condition on the test site(s) i.e. back that can interfere with the reading.
2. Medication which may affect skin response and/or past medical history.
3. Subject having history of diabetes
4. Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.
5. Subject suffering from any active clinically significant skin diseases which may contraindicate.
6. Subject having history of any skin diseases including eczema, atopic dermatitis or active cancer.
7. Participation in any patch test for irritation or sensitization within the last four weeks.
8. Subject having history of asthma or COPD (Chronic obstructive pulmonary disease).
9. Use of any:

   i. Prescribed or over-the-counter (OTC) anti-inflammatory drug within five (5) days prior to application.

   ii. Antihistamine medication or immunosuppressive drugs within seven (7) days prior to first patch application.

   iii. Systemic or topical corticosteroids at patch site within four (4) weeks of test product application (steroidal nose drops and/or eye drops are permitted)
10. Topical drugs used at application site.
11. Subject with Self-reported Immunological disorders such as HIV positive, AIDS and/or systemic lupus erythematous.
12. Individual who has a medical condition or is taking or has taken a medication which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.
13. Subject with known allergy or sensitization to medical adhesives, bandages.
14. Participation in other patch study simultaneously.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the dermatological safety of the test products | Post patch removal of 30 minutes, 24 hours & 168 hours
  Application sites will be evaluated for scoring the reaction, namely, erythema, dryness, and wrinkles on a 0-4 point scale separately for each parameter and oedema as per draize scale

SECONDARY OUTCOMES:
Safety of the skin | At T30 minutes and 24 hours post patch removal. Scoring can be done at T168 hours post-patch removal if required.
  To evaluate the Safety of the skin by visual dermatological assessment by 0: No reaction and 4 Severe Reaction

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Principal Investigator — NovoBliss Research Private Limited
Locations (1):
- NovoBliss Research Private Limited, Ahmedabad, India

IPD SHARING:
Plan to Share IPD: No